CLINICAL TRIAL: NCT06670001
Title: MOtivating Physical Activity With BehaVioral Economics in Heart Failure With Preserved Ejection Fraction (MOVE-HF)
Brief Title: MOVE-HF MOtivating Physical Activity With BehaVioral Economics in Heart Failure With Preserved Ejection Fraction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 855906; 1R01HL174691 (NIH)
Record Dates: First submitted 2024-10-31; First posted 2024-11-01 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: HFpEF - Heart Failure With Preserved Ejection Fraction

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): In addition to using a wearable device, participants in the control arm will receive a daily notification of their step count from the previous day.
- Gamification plus social incentive (Experimental): Participants will receive daily text messages on whether or not they hit their step goal.
  Participants will be entered into a game, that runs for 6 months. Each week they receive 70 points. If the step goal was met they keep their points. If not, they lose 10 points. At the end of the week if they have at least 40 points they move up a level. If not, they drop a level.
  They will receive twice-weekly motivational or educational text messages that highlight the effect of exercise on functional capacity in patients with HFpEF.
  Participants will select a family member or friend who will serve as a support partner. We hold a 3-way phone call with the participant and partner to discuss ways they can help the participant meet their goal. The support partner will receive a weekly email reminding him/her of these approaches and updating him/her on the participant's progress including accumulated points, level in the game, and average step count.
  Interventions: Behavioral: Gamification plus social incentive
- Gamification plus competition (Experimental): Participants will receive daily text messages on whether or not they hit their step goal.
  Participants will be entered into a game, that runs for 6 months. Each week they receive 70 points. If the step goal was met they keep their points. If not, they lose 10 points. At the end of the week if they have at least 40 points they move up a level. If not, they drop a level.
  They will receive twice-weekly motivational or educational text messages that highlight the effect of exercise on functional capacity in patients with HFpEF. Participants will have access to a leaderboard that will include two other participants. Participants will be ranked on the leaderboard by total points over the course of the study. They will receive a weekly text message with their position on the leaderboard.
  Interventions: Behavioral: Gamification plus competition

INTERVENTIONS:
Behavioral: Gamification plus social incentive — Participants in the Gamification plus social incentive intervention arm will receive gamification and social incentives as part of the intervention. See arm descriptions for more detail.
  Arms: Gamification plus social incentive
Behavioral: Gamification plus competition — Participants in the Gamification plus competition intervention arm will receive gamification and a competition as part of the intervention. See arm descriptions for more detail.
  Arms: Gamification plus competition

SUMMARY:
This is a three-arm, randomized, controlled trial to test the effectiveness of gamification plus a social incentive - either social support or competition - to increase adherence to physical activity among individuals with HFpEF. There will be a 2-week run-in period to obtain baseline measures of physical activity, followed by a 6-month intervention period and then a 3-month follow-up period.

DETAILED DESCRIPTION:
Heart failure (HF) with preserved ejection fraction (HFpEF), a syndrome characterized by exercise intolerance due to breathlessness and fatigue, is a major public health problem rising in prevalence. No pharmacologic strategy has been shown to consistently improve functional capacity of HFpEF patients, though exercise training is beneficial. However, reimbursement barriers and access limitations preclude widespread implementation of cardiac rehabilitation. Despite the association between increased physical activity, lower HF hospitalization, and improved quality of life, physical activity levels remain dismally low in HF patients. This is a three-arm, randomized, controlled trial to test the effectiveness of gamification plus a social incentive - either social support or competition - to increase adherence to physical activity among individuals with HFpEF. There will be a 2-week run-in period to obtain baseline measures of physical activity, followed by a 6-month intervention period and then a 3-month follow-up period. All participants will be asked to use the wearable device during the day every day during the intervention and follow-up periods. The three interventions by study arm will vary as follows: Control, Gamification plus social incentive which includes; Pre commitment, support partner, a game using; points, levels, fresh starts, trophies and automated coaching. Competition arm which includes; Pre commitment, a game using; points, levels, fresh starts, trophies and automated coaching and a competition with other participants and access to the leadership board.

ELIGIBILITY:
Inclusion Criteria:

Adults (age ≥ 18 years) who: 1) have a diagnosis of heart failure with preserved ejection; 2) have an ejection fraction ≥ 50%; 3) meet ONE of the following criteria: any history of hospitalization with a primary diagnosis of heart failure with preserved ejection fraction, BNP > 75 pg/mL (> 225 pg/mL in patients with atrial fibrillation), H2FPEF score ≥ 5, OR elevated pulmonary capillary wedge pressure on right heart catheterization (≥ 15 mm Hg at rest or ≥ 25 mm Hg with exercise); 4) own a smartphone or tablet capable of connecting to the internet; 5) are able to read English; 6) are able to provide informed consent

Exclusion Criteria:

Participants will be excluded if they are currently participating in another interventional physical activity study, have medical conditions prohibiting ambulation without assistance (including use of an assistive device other than a cane) or participation in an exercise program, if a 9-month physical activity program is infeasible or unsafe, upcoming cardiovascular procedures (e.g. stent or surgery) or if the patient is at a high level of physical activity (>7500 steps per day) or very low level of physical activity (< 1000 steps/day) at baseline. Patients taking > 7500 steps/day will be excluded based on data showing that increasing step count beyond 7500 steps/day does not improve outcomes in all-comer populations, and to ensure that we are recruiting a population of patients with symptomatic HF. Patients taking < 1000 steps/day at baseline will be excluded to ensure that we will not enroll very frail patients with a need for more intensive exercise training or physical therapy. To ensure that we are capturing patients who are limited in their exertional capacity by heart failure, we will also exclude patients with dementia, end-stage renal disease on dialysis, cirrhosis, cardiac surgery or transcatheter valve replacement within the last year, severe aortic stenosis or severe mitral stenosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2025-06-05 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is the change in mean daily step counts from baseline through the 3-month post-intervention follow-up period. | 9 months
  The primary outcome is the change in mean daily step counts from baseline through the 3-month post-intervention follow-up period.

SECONDARY OUTCOMES:
Change in mean daily steps from baseline to through the 6-month intervention period | 6 months
  Change in mean daily steps from baseline to through the 6-month intervention period
Change in Kansas City Cardiomyopathy Questionnaire-12 (KCCQ-12) score from baseline through the 6-month intervention period | 6 months
  Change in Kansas City Cardiomyopathy Questionnaire-12 (KCCQ-12) score from baseline through the 6-month intervention period
Change in Kansas City Cardiomyopathy Questionnaire-12 (KCCQ-12) score from baseline through the 3-month post-intervention follow-up period | 9 months
  Change in Kansas City Cardiomyopathy Questionnaire-12 (KCCQ-12) score from baseline through the 3-month post-intervention follow-up period
Change in six-minute walk distance from baseline through the 6-month intervention period | 6 months
  Change in six-minute walk distance from baseline through the 6-month intervention period
Change in six-minute walk distance from baseline through the 3-month post-intervention follow-up period | 9 months
  Change in six-minute walk distance from baseline through the 3-month post-intervention follow-up period

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Fanaroff, MD, MHS, Principal Investigator — University of Pennsylvania
Locations (1):
- The University of Pennsylvania, Philadelphia, Pennsylvania, United States